CLINICAL TRIAL: NCT00706979
Title: A Novel Treatment to Boost Quit Attempts and Cessation Among Unmotivated Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA021619-01A1 (NIH); 1R01DA021619-01A1 (NIH)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2010-10

CONDITIONS: Smoking; Smoking Cessation
Keywords: smoking; smoking cessation; nicotine replacement therapy
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Practice Quit Attempt plus Nicotine Replacement Therapy
  Interventions: Other: Practice Quit Attempt plus nicotine lozenge
- 2 (Active Comparator): Practice Quit Attempt only
  Interventions: Behavioral: Practice Quit Attempt only

INTERVENTIONS:
Other: Practice Quit Attempt plus nicotine lozenge — nicotine lozenge, 2 mg or 4 mg
  Other Names: Nicotine lozenge; Nicotine Replacement Therapy (NRT)
  Arms: 1
Behavioral: Practice Quit Attempt only — Practice Quit Attempts (PQA) message aided by brief advice and self-help materials
  Arms: 2

SUMMARY:
A sample of smokers who have no current plans to quit will be recruited for this study and randomized to one of two intervention conditions:

1. Practice Quit Attempt (PQA) aided by brief advice and self-help materials, or
2. PQA aided by advice and self-help materials plus nicotine replacement therapy (NRT).

This study will test whether adding free nicotine replacement therapy to brief advice to undertake a practice quit attempt will motivate more smokers to make a serious attempt to stop smoking than brief advice without NRT. All treatments and assessments will be delivered via telephone and mailing. The primary outcome of interest is the incidence of a serious attempt to permanently stop smoking made over a six-month study period.

Our specific hypotheses are as follows:

Hypothesis 1: Helping smokers to make a practice quit attempt aided by NRT will result in a higher incidence of making a serious effort to quit smoking permanently, compared to an aided practice quit attempt without NRT. We also expect provision of NRT will increase point prevalence abstinence at 6 month follow-up.

Hypothesis 2: This relationship between NRT-aided practice quit attempts and quit behaviors will be mediated by a) increased smoking related self efficacy, b) increased belief in the efficacy of NRT, c) fewer concerns about adverse events of NRT, d) increased social support for not smoking, and e) less withdrawal distress and craving during the practice quit attempt.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker of at least 10 cigarettes per day
* Interested in quitting at some time
* Not currently interested in quitting smoking
* Access to telephone (home or work) for 6 month study period

Exclusion Criteria:

* Monthly cigar, pipe, or smokeless tobacco use
* Current pregnancy or breastfeeding
* Recent cardiovascular distress
* Phenylketonuria (PKU)
* Previous use of nicotine replacement therapy (gum, patch, lozenge, inhaler, or nasal spray)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Carpenter, Ph.D., Principal Investigator — Medical University of South Carolina

REFERENCES:
- [Derived] Carpenter MJ, Hughes JR, Gray KM, Wahlquist AE, Saladin ME, Alberg AJ. Nicotine therapy sampling to induce quit attempts among smokers unmotivated to quit: a randomized clinical trial. Arch Intern Med. 2011 Nov 28;171(21):1901-7. doi: 10.1001/archinternmed.2011.492. PMID 22123796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1/2009 - 2/2010 via the internet from an email database of potential enrollees provided by a market research firm. Eligible participants were mailed an informed consent and asked to return a signed copy if they wished to participate. Research staff then made calls to initiate formal study enrollment.
Pre-assignment Details: Participants were randomized to treatment group in a 1:1 ratio using a random number generator with block randomization before research staff made calls to initiate formal study enrollment.
Groups:
- Practice Quit Attempt Plus Nicotine Replacement Therapy: This group received both the behavioral exercise of a practice quit attempt (PQA) and free nicotine replacement therapy (NRT) in the form of a lozenge for a 6-week treatment period.
- Practice Quit Attempt Only: This group served as the control group and received only the behavioral exercise of a practice quit attempt (PQA).
Period: Overall Study
Arm/Group | Practice Quit Attempt Plus Nicotine Replacement Therapy | Practice Quit Attempt Only
Started | 426 | 423
Completed | 426 | 423
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Practice Quit Attempt Plus Nicotine Replacement Therapy | Practice Quit Attempt Only | Total
Number analyzed (Participants) | 426 | 423 | 849
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 382 | 389 | 771
  >=65 years | 44 | 34 | 78
Age Continuous [Mean (Standard Deviation); unit: years] | 50.5 (11.8) | 50.7 (11.4) | 50.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 279 | 545
  Male | 160 | 144 | 304
Region of Enrollment [Number; unit: participants]
  United States | 426 | 423 | 849

OUTCOME MEASURES:

1. Primary Outcome: A Serious Quit Attempt in Which the Participant Intends to Permanently Stop Smoking
Description: The primary outcome was an attempt to quit smoking for good. To distinguish from a PQA, we specifically asked participants if they tried to quit smoking with the intent of quitting for good. Quit attempts were defined as any self-defined attempt to quit for good.
Time Frame: From study enrollment through six month follow-up
Population: All analyses were based on intent-to-treat approach; participants with missing data were assumed to have not made any quit attempts or quit.
Measure: Number; unit: participants
Arm/Group | Practice Quit Attempt Plus Nicotine Replacement Therapy | Practice Quit Attempt Only
Number analyzed (Participants) | 426 | 423
participants | 208 | 168
Statistical Analysis 1: Comparison: Practice Quit Attempt Plus Nicotine Replacement Therapy vs Practice Quit Attempt Only; A logistic regression model was used to examine the primary hypothesis that NRT-enhanced PQAs would yield a higher rate of any ever-occurring quit attempt; Test type: Superiority or Other; p = 0.008, Regression, Logistic; Risk Ratio (RR) = 1.2, 95% CI 2-sided [1.1 to 1.4]

2. Secondary Outcome: Abstinence From Cigarette Smoking, Where Abstinence is Defined as Self-report of Not Smoking at All for 7 Consecutive Days
Time Frame: At any point during the study
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Practice Quit Attempt Plus Nicotine Replacement Therapy | Practice Quit Attempt Only
Number analyzed (Participants) | 426 | 423
participants | 82 | 63
Statistical Analysis 1: Comparison: Practice Quit Attempt Plus Nicotine Replacement Therapy vs Practice Quit Attempt Only; A logistic regression model was used to examine the secondary hypothesis that NRT-enhanced PQAs would yield a higher rate of 7 days of abstinence at some point during the study; Test type: Superiority or Other; p = 0.09, Regression, Logistic; Risk Ratio (RR) = 1.3, 95% CI 2-sided [1.0 to 1.7]

3. Primary Outcome: A 24 Hour Serious Quit Attempt in Which the Participant Intends to Permanently Stop Smoking
Description: Serious quit attempt of >=24hrs, which fits the CDC's definition of a quit attempt.
Time Frame: From study enrollment through six month follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Practice Quit Attempt Plus Nicotine Replacement Therapy | Practice Quit Attempt Only
Number analyzed (Participants) | 426 | 423
participants | 185 | 143
Statistical Analysis 1: Comparison: Practice Quit Attempt Plus Nicotine Replacement Therapy vs Practice Quit Attempt Only; A logistic regression model was used to examine the primary hypothesis that NRT-enhanced PQAs would yield a higher rate for the primary outcome of any 24hr quit attempt; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Risk Ratio (RR) = 1.3, 95% CI 2-sided [1.1 to 1.5]

4. Secondary Outcome: Abstinence From Cigarette Smoking, Where Abstinence is Defined as Self-report of Not Smoking at All for 7 Consecutive Days
Time Frame: At 6-month follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Practice Quit Attempt Plus Nicotine Replacement Therapy | Practice Quit Attempt Only
Number analyzed (Participants) | 426 | 423
participants | 68 | 57
Statistical Analysis 1: Comparison: Practice Quit Attempt Plus Nicotine Replacement Therapy vs Practice Quit Attempt Only; A logistic regression model was used to examine the secondary hypothesis that NRT-enhanced PQAs would yield a higher rate for 7 days of abstinence at the six month follow-up; Test type: Superiority or Other; p = 0.3, Regression, Logistic; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.9 to 1.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected in the Practice Quit Attempt (PQA) + Nicotine Replacement Therapy (NRT) group only. They were collected at every follow-up study visit, which included 5 time points over a 7.5 month (32 weeks) period.
Arm/Group | Practice Quit Attempt Plus Nicotine Replacement Therapy | Practice Quit Attempt Only
Serious Adverse Events (participants affected / at risk) | 0/426 | 1/423
Other Adverse Events (participants affected / at risk) | 179/426 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Practice Quit Attempt Plus Nicotine Replacement Therapy (N=426) | Practice Quit Attempt Only (N=423)
Death (Renal and urinary disorders) | 0 (0) | 1 (1) — We were notified of the death of a participant from bladder cancer in the control group(PQA Only group, did not receive nicotine replacement therapy) by the participant's wife.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Practice Quit Attempt Plus Nicotine Replacement Therapy (N=426) | Practice Quit Attempt Only (N=0)
Nausea/stomach upset (dyspepsia) (Gastrointestinal disorders) | 80 (80) | 0 (0)
Throat irritation (General disorders) | 60 (60) | 0 (0)
Hiccups (General disorders) | 45 (45) | 0 (0)
Heartburn (Gastrointestinal disorders) | 23 (23) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No